CLINICAL TRIAL: NCT02417415
Title: Local Heat Stress in Autonomic Failure Patients With Supine Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University (Other)
Responsible Party: Principal Investigator, Italo Biaggioni, Professor of Medicine, Vanderbilt University
Organization: Vanderbilt University Medical Center (Other)
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Other
Other Study IDs: 141523
Record Dates: First submitted 2015-04-10; First posted 2015-04-15 (Estimated); Results first posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2021-12

CONDITIONS: Hypertension; Pure Autonomic Failure; Multiple System Atrophy; Autonomic Failure
Keywords: Supine hypertension; Autonomic failure; Heat intolerance; Orthostatic hypotension; Heat stress
MeSH Terms: conditions — Hypertension; Pure Autonomic Failure; Multiple System Atrophy; Hypotension, Orthostatic; Heat Stress Disorders | interventions — salicylhydroxamic acid

STUDY DESIGN:
Intervention Model Description: randomized, 2-arm crossover study (heat vs. sham)
Who Masked: Participant
Masking Description: Patients were blinded to the intervention
Oversight: Data Monitoring Committee: No

ARMS (2):
- Local Heat Stress (Experimental): Passive heat-stress using a commercial heating pad applied over the abdomen and part of the torso
  Interventions: Other: Passive heat stress
- Control (Non-heating) (Sham Comparator): Commercial heating pad applied over the abdomen and part of the torso but turned off
  Interventions: Other: Control (non-heating)

INTERVENTIONS:
Other: Passive heat stress — Passive heat stress will be applied with a commercial heating pad that covers all the abdomen and part of the torso to provide local heating at ~44ºC continuously for 2 hr.
  Other Names: Heating pad
  Arms: Local Heat Stress
Other: Control (non-heating) — Heating pad will be applied over the abdomen and part of the torso but it will be turned off.
  Other Names: sham
  Arms: Control (Non-heating)

SUMMARY:
Patients with autonomic failure are characterized by disabling orthostatic hypotension (low blood pressure on standing), and at least half of them also have high blood pressure while lying down (supine hypertension). Exposure to heat, such as in hot environments, often worsens their orthostatic hypotension. The causes of this are not fully understood. The purpose of this study is to evaluate whether applying local heat over the abdomen of patients with autonomic failure and supine hypertension would decrease their high blood pressure while lying down. This will help us better understand the mechanisms underlying this phenomenon, and may be of use in the treatment of supine hypertension.

DETAILED DESCRIPTION:
Primary autonomic failure is a neurodegenerative condition characterized by severe impairment of the autonomic nervous system. The clinical hallmark of autonomic failure is disabling orthostatic hypotension, but at least half of patients are also hypertensive while lying down. This supine hypertension can be severe and associated with end-organ damage and worsening of orthostatic hypotension due to increased pressure natriuresis. It also complicates the management of these patients by limiting the use of daytime pressor agents for the treatment of orthostatic hypotension.

It is well known that heat exposure (e.g. hot weather or a hot bath or shower) produces an acute and temporary worsening of orthostatic hypotension in autonomic failure patients. However, the mechanisms underlying this phenomenon are completely unexplored. Factors that may predispose autonomic failure patients to the acute lowering blood pressure effects of heat stress include 1) impaired heat dissipation due to inability to sweat, 2) preserved heat-mediated skin vasodilation, and 3) blunted sympathetic hemodynamic responses to maintain blood pressure. In this study, we test the hypothesis that moderate levels of local (abdominal) passive heat stress will lower blood pressure in autonomic failure patients with supine hypertension.

To test this hypothesis, we propose this pilot study with the following specific aims:

1. To evaluate the acute blood pressure effects of local passive heat stress in autonomic failure patients with supine hypertension, we will compare changes in BP between controlled local heat stress (~44ºC) using a commercial heating pad that covers the abdomen and part of the torso, and a control (non-heating) study day using the same heating pad but turned off.
2. To evaluate the mechanisms underlying BP changes during local heat stress, we will compare changes in hemodynamic parameters (cardiac output, stroke volume and peripheral vascular resistance), segmental fluid shifts (measured by segmental bioimpedance), skin blood flow and skin temperature between the heat and non-heating study days.

ELIGIBILITY:
Inclusion Criteria:

* Male and female patients, between 18-80 yrs., with primary autonomic failure (Parkinson Disease, Multiple System Atrophy, and Pure Autonomic Failure) and supine hypertension. Supine hypertension will be defined as SBP≥150 mmHg.
* Patients able and willing to provide informed consent.

Exclusion Criteria:

* Pregnancy
* Significant cardiac, renal or hepatic illness, or with contraindications to administration of pressor agents or with other factors, which in the investigator's opinion would prevent the subject from completing the protocol including clinically significant abnormalities in clinical, mental or laboratory testing.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 22 (Actual)
Dates: Start 2015-04 (Actual); Primary Completion 2021-02 (Actual); Study Completion 2021-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Italo Biaggioni, MD, Principal Investigator — Vanderbilt University
Locations (1):
- Vanderbilt University, Nashville, Tennessee, United States

REFERENCES:
- [Derived] Okamoto LE, Celedonio JE, Smith EC, Gamboa A, Shibao CA, Diedrich A, Paranjape SY, Black BK, Muldowney JAS 3rd, Peltier AC, Habermann R, Crandall CG, Biaggioni I. Local Passive Heat for the Treatment of Hypertension in Autonomic Failure. J Am Heart Assoc. 2021 Apr 6;10(7):e018979. doi: 10.1161/JAHA.120.018979. Epub 2021 Mar 19. PMID 33739123

RESULTS

PARTICIPANT FLOW:
Groups:
- Local Heat Stress Then Sham Control: Passive heat-stress of 40-42 degrees applied with an electric heating pad over the abdomen and part of the torso for up to 2 hours on study day 1 and sham control (heating pad turned off for up to 2 hours) on study day 2
- Sham Control Then Local Heat Stress: Sham control (heating pad turned off for up to 2 hours) on study day 1 and local heat stress of 40-42 degrees applied with an electric heating pad over the abdomen and part of the torso for up to 2 hours on study day 2.
Period: Overall Study
Arm/Group | Local Heat Stress Then Sham Control | Sham Control Then Local Heat Stress
Started | 13 | 9
Completed | 13 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- All Study Participants: Participants who were randomized to receive local passive heat stress and sham control in any order.
Arm/Group | All Study Participants
Number analyzed (Participants) | 22
Age, Continuous [Mean (Standard Deviation); unit: years] | 73 (6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6
  Male | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 21
  More than one race | 0
  Unknown or Not Reported | 0
BMI [Mean (Standard Deviation); unit: kg/m^2] | 27 (4)
Disease Duration [Mean (Standard Deviation); unit: years] | 7 (4)
Diagnosis [Count of Participants; unit: Participants]
  Pure Autonomic Failure | 14
  Parkinson Disease + Autonomic Failure | 7
  Multiple System Atrophy | 1
Medical history of essential hypertension [Count of Participants; unit: Participants] | 10
Heat intolerance [Count of Participants; unit: Participants] | 15
Systolic BP, supine [Mean (Standard Deviation); unit: mm Hg] | 170 (23)
Systolic BP, upright [Mean (Standard Deviation); unit: mm Hg] | 100 (33)
Heart rate, supine [Mean (Standard Deviation); unit: bpm] | 67 (12)
Heart rate, upright [Mean (Standard Deviation); unit: bpm] | 77 (11)
Plasma norepinephrine, supine [Mean (Standard Deviation); unit: pg/mL] — Population: Blood samples could not be obtained in 3 subjects
  pg/mL
    number analyzed (Participants) | 19
    (all) | 132 (70)
Plasma norepinephrine, upright [Mean (Standard Deviation); unit: pg/mL] — Population: Blood samples could not be obtained in 2 subjects
  pg/mL
    number analyzed (Participants) | 20
    (all) | 199 (136)

OUTCOME MEASURES:

1. Primary Outcome: Change in Systolic Blood Pressure
Description: Change from baseline in systolic blood pressure at 2 hr post-intervention
Time Frame: 2 hours of heat stress or sham
Measure: Mean (Standard Error); unit: mm Hg
Groups:
- Local Heat Stress: Passive heat-stress using a commercial heating pad applied over the abdomen and part of the torso
  Passive heat stress: Passive heat stress was applied with a commercial heating pad that covers all the abdomen and part of the torso to provide local heating at 40-42 degrees continuously for 2 hr.
- Control (Non-heating): Commercial heating pad applied over the abdomen and part of the torso but turned off
  Control (non-heating): Heating pad was applied over the abdomen and part of the torso but it will be turned off for up to 2 hours
Arm/Group | Local Heat Stress | Control (Non-heating)
Number analyzed (Participants) | 22 | 22
mm Hg | 19 (4) | 3 (4)

2. Secondary Outcome: Percent Change in Hemodynamic Parameters (Cardiac Output, Stroke Volume and Systemic Vascular Resistance)
Description: Percent change from baseline ([post-intervention - baseline]/baseline X 100) in cardiac output, stroke volume and systemic vascular resistance at 2 hours post-intervention
Time Frame: 2 hours of heat stress or sham
Population: Systemic hemodynamics were measured in 13 of the 22 participants
Measure: Mean (Standard Error); unit: percentage change
Arm/Group | Local Heat Stress | Control (Non-heating)
Number analyzed (Participants) | 13 | 13
percentage change
  Cardiac Output | -15 (5) | -2 (4)
  Stroke Volume | -18 (5) | -4 (4)
  Systemic Vascular Resistance | 9 (6) | 4 (5)

ADVERSE EVENTS:
Time Frame: Adverse event information was collected for all interventions every 20 to 30 minutes for up to 2.5 hours.
Arm/Group | Local Heat Stress | Control (Non-heating)
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/22
Other Adverse Events (participants affected / at risk) | 0/22 | 0/22

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-09-13): https://cdn.clinicaltrials.gov/large-docs/15/NCT02417415/Prot_SAP_000.pdf